CLINICAL TRIAL: NCT06877845
Title: Effects of Postural Corrector and Activity Tracker for Enhanced Post-operative Rehabilitation of Total Knee Replacement
Brief Title: Postural Correctors & Activity Trackers in Total Knee Replacement Rehab
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REC-01006 Nauman Nazir
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-03

CONDITIONS: Total Knee Replacement
Keywords: Pain; Knee Function; Post-operative Rehabilitation
MeSH Terms: conditions — Pain | interventions — Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activity Tracker & Postural Corrector (Experimental): Activity Tracker & Postural Corrector
  along with conventional treatment
  Interventions: Other: Activity Tracker & Postural Corrector; Other: Conventional Therapy
- Conventional Treatment (Active Comparator): * HOT PACKS:for 15 minutes
  * TENS (transcutaneous electric nerve stimulator): for 10 minutes
  * ROMs(range of motions): at knee joint Passive and Active-Assisted Knee Flexion and Extension Quadriceps Sets Straight Leg Raises (SLR) Ankle Pumps
  * Strengthening Exercises: Quadriceps Strengthening, Hamstring Curls, Gluteal Strengthening & Calf Raises
  Total Duration of Exercise Session: 25 minutes
  Interventions: Other: Conventional Therapy

INTERVENTIONS:
Other: Activity Tracker & Postural Corrector — Use of Activity Tracker & Postural Corrector along with following baseline treatment.
  * HOT PACKS:for 15 minutes
  * TENS (transcutaneous electric nerve stimulator): for 10 minutes
  * ROMs(range of motions): at knee joint Passive and Active-Assisted Knee Flexion and Extension Quadriceps Sets Straight Leg Raises (SLR) Ankle Pumps
  * Strengthening Exercises:
  Quadriceps Strengthening Hamstring Curls Gluteal Strengthening Calf Raises
  Total Duration of Exercise Session: 25 minutes
  Arms: Activity Tracker & Postural Corrector
Other: Conventional Therapy — * HOT PACKS:for 15 minutes
  * TENS (transcutaneous electric nerve stimulator): for 10 minutes
  * ROMs(range of motions): at knee joint Passive and Active-Assisted Knee Flexion and Extension Quadriceps Sets Straight Leg Raises (SLR) Ankle Pumps
  * Strengthening Exercises:
  Quadriceps Strengthening Hamstring Curls Gluteal Strengthening Calf Raises
  Total Duration of Exercise Session: 25 minutes

SUMMARY:
* To assess the impact of postural corrector on post-operative knee function and activity
* To evaluate the role of activity tracker in monitoring and enhancing post-operative rehabilitation
* To assess the effects of postural corrector and activity tracker on pain management during rehabilitation

DETAILED DESCRIPTION:
Knee osteoarthritis is a major public health threat. Chronic pain and incapacity related to knee degenerative arthritis (OA) is current among the older population in several developed countries and also the condition is marked by many pathological characteristics, like joint house narrowing and also the formation of osteophytes, Despite the pressing want for effective hindrance and treatment methods, there's a scarcity of comprehensive demographic knowledge on the general prevalence of the un wellness and also the specific subgroups affected

ELIGIBILITY:
Inclusion Criteria:

* Participants who fall in this category will be included in the study.

  * Commercially available devices
  * Post-operative total knee replacement
  * Males and females
  * Age 40 to 60 years

Exclusion Criteria:

* Participants who fall in this category will be excluded from the study.

  * Non wearable devices
  * Patient had been through surgery more than 1 month
  * Patients with any other disorder or disease

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
OKS (Oxford Knee Score) to assess Function and Pain in Knee | 12 Weeks
  The OKS is a patient-reported outcome measure that is used to assess the severity of a knee problem and the effect of knee conditions on a person's life. The questionnaire has 12 questions about pain, function, and limitations in activities, and it provides doctors insight into how much a patient's knee problems are limiting daily activities. You sum the scores for all 12 questions. The scores ranges from zero to 48, zero meaning worst knee function and 48 meaning best knee function.
UCLA Activity Scale for assessing the Physical Activity Level of patients undergoing Knee & Hip Arthoplasty | 12 Weeks
  The UCLA Activity Scale (UCLA) is a questionnaire used to assess physical activity levels in patients undergoing hip or knee arthroplasty, ranging from 1 (low) to 10 (high), and is valuable for measuring changes in self-reported physical activity.
EQ-5D-5L (EuroQol 5-DIMENSION 5-Level) to measure the health-related quality of life (HRQoL) | 12 Weeks
  One popular instrument for evaluating people's health-related quality of life (HRQoL) is the EQ-5D questionnaire. The EQ-5D-5L comprises a VAS in addition to the descriptive system and index score. The VAS asks the responder to rate their general health on a scale of 0 to 100, where 100 is the best possible health and 0 is the worst possible health.
NPRS (NUMERIC PAIN RATING SCALE) for Pain | 12 Weeks
  A straightforward and widely used instrument for determining the degree of pain is the NPRS (Numeric Pain Rating Scale). the NPRS is used to gauge the degree of either acute or chronic pain. Using a 0-10 scale, the NPRS allows users to rate the intensity of their pain by choosing the number that most accurately represents their current level of discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Sadiq, MSPT (OMPT), Principal Investigator — Riphah International University
Locations (1):
- Helping Hand Institute of Rehabilitation Sciences (HHIRS), Mānsehra, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No